CLINICAL TRIAL: NCT04733833
Title: A Randomized, Controlled Study to Evaluate the Efficacy and Safety of VB-201 in Patients With COVID-19
Brief Title: A Study to Evaluate the Efficacy and Safety of VB-201 in Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VB-201-019
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2021-01

CONDITIONS: Severe COVID-19
Keywords: COVID-19; Severe
MeSH Terms: conditions — COVID-19; Lymphoma, Follicular | interventions — 1-palmityl-2-(4-carboxybutyl)-sn-glycero-3-phosphocholine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): VB-201 + standard of care
  Interventions: Drug: VB-201 + Standard of care
- Arm 2 (Active Comparator): Standard of care
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: VB-201 + Standard of care — Daily oral administration of VB-201- 160 mg (80 mg BID) with standard of care
  Arms: Arm 1
Drug: Standard of care — Standard of care
  Arms: Arm 2

SUMMARY:
The purpose of this Phase 2 study is to test safety, efficacy, and tolerability of an oral preparation of VB-201 in patients with severe COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. Signed and approved informed consent before initiation of protocol-specified procedures;
2. Male or female subjects, ≥18 to ≤80 years of age with COVID-19
3. SARS-2-CoV-2 infection confirmed by PCR in the last 8 days
4. Hospitalized
5. Symptoms of Severe COVID-19 as demonstrated by one of the following:

   * Respiratory frequency >30 breaths per minute
   * SpO2 <94% on room air at sea level
   * Ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mmHg
   * lung infiltrates >50%
6. For a female subject; either:

   * subject is of non-childbearing potential, defined as: menopause with amenorrhea >1 years, hysterectomy, or bilateral oopherectomy or
   * agrees to continue to use highly effective methods of birth control defined as those alone or in combination that result in a low failure rate (<1%) when used consistently and correctly throughout the study and for at least one month following treatment termination and have a negative pregnancy test at screening and before the first dose of study drug; Males must use at least one method of contraception (e.g. condom) throughout the study and for 90 days following the last dose of study drug;
7. In the opinion of the investigator, the subject will be compliant and have a high probability of completing the study and all required procedures.

Exclusion Criteria:

1. Evidence of critical COVID-19 based on any of the following

   * Admission to ICU
   * Assisted ventilation (invasive or non-invasive)
   * ECMO or hemofiltration required
   * ARDS
   * Shock
   * Acute Cardiac Failure
2. Dementia
3. Bacterial co-infection
4. Co-infection with other common viral pneumonias (e.g. Influenza)
5. Participation in another interventional clinical trial or intention to participate in another interventional study during the course of this study;
6. In the opinion of the investigator, unlikely to survive for at least 48 hours from screening or anticipate mechanical ventilation within 48 hours
7. Unable to take oral medication
8. History of gastrointestinal illness that may cause nausea and vomiting
9. Subjects with any laboratory test at screening that common medical practice would deem as significantly abnormal. For example:

   * Alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase >5.0 times the upper limit of normal (ULN) or
   * Creatinine clearance <30 mL/min
10. The subject has a known allergy or sensitivity to the study treatment or to any of the excipients contained in the study drug formulation (see list of ingredients in the Investigator's Brochure);
11. Female subject with a positive pregnancy test or nursing, or planning a pregnancy during the course of the study;
12. Unwilling or unable to comply with study requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of VB-201 | Subjects will participate in the study for approximately 7 weeks: up to 1 day for screening and establishment of baseline, followed by 14 days of treatment and a follow-up visit 4 weeks after last dose of study medication.
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 (Time frame: Adverse events will be collected from the time the informed consent is signed through 28 days after the subject's last dose. All adverse events that are ongoing at the time of completion/discontinuation will be followed until resolution or the event is chronic or stable in the opinion of the investigator).

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel